CLINICAL TRIAL: NCT00234117
Title: Overall Assessment of Improvement in Bronchial Asthma Patients With Extraesophageal Reflux After Effective Acid Suppression
Brief Title: Improvement in Bronchial Asthma in Patients With Extraesophageal Reflux After Acid Suppression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ponce Gastroenterology Research (Other)
Collaborators: PriCara, Unit of Ortho-McNeil, Inc. (Industry)
Responsible Party: Dr. Nilda Santiago, Ponce Gastroenterology
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAB-EMR-4037
Record Dates: First submitted 2005-10-05; First posted 2005-10-06 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2005-10

CONDITIONS: Bronchial Asthma; Gastroesophageal Reflux
MeSH Terms: conditions — Asthma; Gastroesophageal Reflux | interventions — Rabeprazole

INTERVENTIONS:
Drug: Rabeprazole

SUMMARY:
The purpose of this study is to determine if 20mg BID of Rabeprazole is effective in controlling GERD in patients with concomitant bronchial asthma and to assess improvement in asthma after reflux control.

DETAILED DESCRIPTION:
Gastroesophageal Reflux Disease has been considered as having a role in the course of asthma, as shown by the improvement of symptoms with adequate acid suppression therapy. It is important to consider and establish the presence of GERD in patients with asthma specially, those who fail to respond to conventional asthma management. It is believed that two mechanisms may play a role in the association between Bronchial Asthma and GERD, most commonly microaspiration of acid causing bronchoconstriction, the second being increased vagal tone.

Establishing an adequate and timely diagnosis and confirming or excluding a relationship between the two entities in asthmatic patients is the first step towards effective patient management. The next important consideration is establishing the correct acid suppression therapy and monitoring response to therapy with objective testing such as Pulmonary Function Testing (PFT) and esophageal pH testing. Since there is not a real "normal" or physiologic reflux measure for patients with extresophageal manifestations as seen in patients with "classic" reflux where a total time of exposure to acid (pH < 4) less than 5% is considered normal, in these patients it will be necessary to establish a more strict pH control than in those with classic GERD. Achieving complete acid control in this population is expected to require higher doses of medication than those used in patients with classic reflux and no extraesophageal manifestations. Thus we have developed this study in which we will assess the response to 20 mg BID dosing of Rabeprazole measured by pH monitoring and then follow improvement in Pulmonary Function Testing ( objective measure),as well as symptomatic response.

ELIGIBILITY:
Inclusion Criteria:

* Moderate Persistent or moderate severe bronchial asthma as determined by the study pulmonologist
* Gastroesophageal Reflux disease

Exclusion Criteria:

* History of hypersensitivity to rabeprazole or its metabolites

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2005-07

PRIMARY OUTCOMES:
Efficacy of rabeprazole treatment will be described using the proportion of the subjects with complete acid suppression at week 12

CONTACTS AND LOCATIONS:
Overall Officials: Alvaro Reymunde, MD, Principal Investigator — Ponce Gastroenterology Research
Locations (1):
- Ponce Gastroentrology Research, Ponce, Puerto Rico